CLINICAL TRIAL: NCT04673747
Title: Intraoperative Manual Correction of Iliosacral Displacement of the Sacroiliac Joint in Total Hip Arthroplasty
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: I.M. Sechenov First Moscow State Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1381
Record Dates: First submitted 2020-12-03; First posted 2020-12-17 (Actual); Last update posted 2021-06-16 (Actual); Status verified 2020-11

CONDITIONS: Total Hip Arthroplasty
Keywords: hip joint; the sacroiliac joint; Iliosacral displacement; manual correction
MeSH Terms: interventions — Arthroplasty, Replacement, Hip

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Total Hip Arthroplasty with intraoperative manual correction) (Experimental): Patients will undergo total hip arthroplasty with intraoperative manual correction of Iliosacral displacement of the sacroiliac joint
  Interventions: Procedure: Total Hip Arthroplasty; Procedure: Manual correction of the sacroiliac joint
- Group 2 (Total hip Arthroplasty: standard method) (Active Comparator): Patients will undergo total hip arthroplasty according to the standard method
  Interventions: Procedure: Total Hip Arthroplasty

INTERVENTIONS:
Procedure: Total Hip Arthroplasty — Total replacement of the head, femoral neck and acetabulum of the hip joint with specialized implants
Procedure: Manual correction of the sacroiliac joint — Manual correction of the iliosacral displacement of the sacroiliac joint in total hip arthroplasty is performed in the operating room after anesthesia just before total hip arthroplasty. It is carried out according to the methodology developed by us.
  Arms: Group 1 (Total Hip Arthroplasty with intraoperative manual correction)

SUMMARY:
Degenerative changes in the hip joint, which are indications for operative treatment, are observed in more than 30% over the age of 50. In most cases, the development of a degenerative process in the hip joint is accompanied by changes in the sacroiliac joint. To improve the quality of life, relieve pain, improve the clinical outcomes of rehabilitation after total hip arthroplasty (THA), an integrated approach to treatment is required.

The investigators have developed a technique for intraoperative manual correction of the ileosacral displacement of the sacroiliac joint during THA. This clinical study compares the use of this technique during THA and THA by standard method.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent of the patient to participate in the study
* Patients with osteoarthritis of the hip joint.
* The opportunity for observation during the entire study period (12 months)
* Mental adequacy, ability, willingness to cooperate and follow the doctor's recommendations

Exclusion Criteria:

* The refusal of a patient from surgery
* The presence of contraindications to surgery
* Severe forms of diabetes (glycosylated hemoglobin >9%)
* Previously performed surgeries on the lumbar spine
* Blood diseases (thrombopenia, thrombocytopenia, anemia with Hb< 90g\l)
* The unwillingness of the patient to conscious cooperation.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2017-06-01 (Actual); Primary Completion 2022-05 (Estimated); Study Completion 2022-05 (Estimated)

PRIMARY OUTCOMES:
Pain assessment | before surgery
  Visual Analogue Scale (VAS) - assessment or the severity of pain syndrome. The score is determined by measuring the distance (mm) on a 10 cm line between the no pain anchor point and the patient's mark, giving a value range from 0 to 100 (0 - min; 100- max)
Pain assessment | 3 months after surgery
  Visual Analogue Scale (VAS) - assessment or the severity of pain syndrome. The score is determined by measuring the distance (mm) on a 10 cm line between the no pain anchor point and the patient's mark, giving a value range from 0 to 100 (0 - min; 100- max)
Pain assessment | 6 months after surgery
  Visual Analogue Scale (VAS) - assessment or the severity of pain syndrome. The score is determined by measuring the distance (mm) on a 10 cm line between the no pain anchor point and the patient's mark, giving a value range from 0 to 100 (0 - min; 100- max)
Pain assessment | 12 months after surgery
  Visual Analogue Scale (VAS) - assessment or the severity of pain syndrome. The score is determined by measuring the distance (mm) on a 10 cm line between the no pain anchor point and the patient's mark, giving a value range from 0 to 100 (0 - min; 100- max)
Hip function assessment | before surgery
  The Harris Hip Score (HSS). The HHS is a measure of disfunction so the higher the score, the better the outcome for the individual. Results can be recorded and calculated online. The maximum score possible is 100. Results can be interpreted with the following: <70 = poor result; 70-80 = fair, 80-90 = good, and 90-100 = excellent.
Hip function assessment | 3 months after surgery
  The Harris Hip Score (HSS). The HHS is a measure of disfunction so the higher the score, the better the outcome for the individual. Results can be recorded and calculated online. The maximum score possible is 100. Results can be interpreted with the following: <70 = poor result; 70-80 = fair, 80-90 = good, and 90-100 = excellent.
Hip function assessment | 6 months after surgery
  The Harris Hip Score (HSS). The HHS is a measure of disfunction so the higher the score, the better the outcome for the individual. Results can be recorded and calculated online. The maximum score possible is 100. Results can be interpreted with the following: <70 = poor result; 70-80 = fair, 80-90 = good, and 90-100 = excellent.
Hip function assessment | 12 months after surgery
  The Harris Hip Score (HSS). The HHS is a measure of disfunction so the higher the score, the better the outcome for the individual. Results can be recorded and calculated online. The maximum score possible is 100. Results can be interpreted with the following: <70 = poor result; 70-80 = fair, 80-90 = good, and 90-100 = excellent.

CONTACTS AND LOCATIONS:
Overall Officials: Alexey Lychagin, MD, Phd, Study Chair — IM Sechenov University
Locations (1):
- Sechenov University, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Alexey L, Vadim C, Marina L, Evgenia T, Kseniya Y, Roza YH, Alexey K, Ivan V. Prognostic role of affected side of the sacroiliac joint in pain recurrence after total hip arthroplasty with prior manual correction of iliosacral dislocation: prospective randomized clinical study. Int Orthop. 2022 Mar;46(3):541-548. doi: 10.1007/s00264-021-05240-w. Epub 2021 Oct 16. PMID 34655319